CLINICAL TRIAL: NCT04149509
Title: ACT NOW Longitudinal Study: Outcomes of Babies With Opioid Exposure Study
Acronym: OBOE
Status: Active, not recruiting | Type: Observational
Sponsor: Advancing Clinical Trials in Neonatal Opioid Withdrawal (ACT NOW) Program (Network)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: ACTNOW-03; 1PL1HD101059-01 (NIH); RL1HD104251 (NIH); RL1HD104252 (NIH); RL1HD104253 (NIH); RL1HD104254 (NIH)
Record Dates: First submitted 2019-10-24; First posted 2019-11-04 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Neonatal Opioid Withdrawal Syndrome
Keywords: NOWS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposed: Infants born ≥ 37 weeks gestation with second or third trimester opioid exposure as determined by maternal urine toxicology screen at delivery; maternal history; and/or infant urine, meconium, or umbilical cord toxicology screen.
- Unexposed - Controls: Infants born ≥ 37 weeks gestation with no antenatal drug exposure as determined by maternal urine toxicology screen at delivery and/or maternal history. We will match control infants to exposed infants based on Clinical Site and up to 60 days after the date of birth of the exposed infant , recruiting 1 control for every other exposed infant at each site.

SUMMARY:
The objective of this longitudinal cohort study is to quantify the effects of antenatal opioid exposure on the trajectory of brain development over the first 2 years of life, examine associations with developmental and neurobehavioral outcomes, and explore how specific factors (differing antenatal and postnatal exposures, severity of neonatal opioid withdrawal, maternal stress/depression/parenting) modify these effects

DETAILED DESCRIPTION:
This objective of this longitudinal cohort study is to prospectively examine the medical, neuroanatomical, neurodevelopmental, behavioral, and social/family/home outcomes of infants who were exposed to opioids in utero. Match control infants will be recruited into the study and based on birth hospital and birth month of the exposed infants. The study will quantify the effects of antenatal opioid exposure on the trajectory of brain development over the first 2 years of life, examine associations with developmental and neurobehavioral outcomes, and explore how specific factors (differing antenatal and postnatal exposures, severity of neonatal opioid withdrawal, maternal stress/depression/parenting) modify these effects. The investigators hypothesize that neural connectivity and neuroanatomical volumes are altered by antenatal opioid exposure and that the magnitude of these alterations correlates with developmental and behavioral outcomes. Further, maternal and environmental factors interact with antenatal opioid exposure to influence the trajectories of connectivity, development, and behavior over the first 2 years of life.

ELIGIBILITY:
Inclusion Criteria:

* Exposed infants: Born ≥37 weeks gestation with second or third trimester opioid exposure
* Control infants: Born ≥37 weeks gestation with no antenatal drug exposure

Exclusion Criteria:

1. Infants with known chromosomal or congenital anomalies potentially affecting the central nervous system
2. Apgar score at 5 minutes of <5
3. Any requirement for positive pressure ventilation in the NICU
4. Inability to return for outpatient MRI and/or follow-up
5. IUGR <3rd percentile
6. Heavy alcohol use during pregnancy (8+ drinks per week).

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants will be prescreened at participating birth hospitals using the inclusion and exclusion criteria listed below.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome related to brain development: White Matter Volume | Birth to 22-24 months of age
  Volumetric analysis will be done with the white matter volume obtained from each of the MRI images collected from birth until 22-24 months of age. The differences between the exposed and non-exposed groups will be calculated.
Primary outcome related to brain development: Cortical Gray Matter Volume | Birth to 22-24 months of age
  Volumetric analysis will be done with the cortical gray matter volume obtained from each of the MRI images collected from birth until 22-24 months of age. The differences between the exposed and non-exposed groups will be calculated.
Primary outcome related to brain development: Deep Gray Matter Volume | Birth to 22-24 months of age
  Volumetric analysis will be done with the deep gray matter volume obtained from each of the MRI images collected from birth until 22-24 months of age. The differences between the exposed and non-exposed groups will be calculated.
Primary outcome related to brain development: Lateral Ventricle Volume | Birth to 22-24 months of age
  Volumetric analysis will be done with the lateral ventricle volume obtained from each of the MRI images collected from birth until 22-24 months of age. The differences between the exposed and non-exposed groups will be calculated.
Primary outcome related to brain development: External cerebrospinal fluid | Birth to 22-24 months of age
  Volumetric analysis will be done with the external cerebrospinal fluid volume obtained from each of the MRI images collected from birth until 22-24 months of age. The differences between the exposed and non-exposed groups will be calculated.
Primary outcome related to behavioral and development: Bayley Scales of Infant Development | 22-24 months of age
  The Bayley Scales of Infant Development is considered the gold standard assessment of early child development and includes cognitive, language, fine motor, and gross motor subscales. Subscale scores each range from 1 - 19, with higher scores indicating higher performance.
Primary outcome related to behavioral and development: Spot Vision Screener | 22-24 months of age
  The vision screener and auto-refractor detects amblyopia risk factors such as myopia, hyperopia, astigmatism, anisometropia, gaze, and anisocoria. Results are reported as "all measurements in range-pass" or "complete eye exam recommended-fail" based on manufacturer criteria for age. If the screen recommends a complete eye exam, the reason for failure (of the 6 factors listed above) and affected eye(s) will be recorded.
Primary outcome related to behavioral and development: BITSEA | 22-24 months of age
  Brief Infant-Toddler Social and Emotional Assessment (BITSEA) is a 42 item tool that is useful for identifying social-emotional problems and/or deficits in children. BITSEA includes the following subscales: Competence (11 Items, min score:0, max score:22), problem behaviors--dysregulation (8 items, min score:0, max score:16) , externalizing (6 items, min score:0, max score:12), internalizing (8 items, min score:0, max score:16), Autism Spectrum Disorder (17 Items, min score:0, max score:34), and Red Flags (14 items, min score:0, max score:28).The questions overlap and the problem subscale is a combination of dysregulation, externalizing, and internalizing. Higher problem scores indicate greater levels of social-emotional/behavioral problems. Lower Competence scores indicate possible delay/deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Bann, PhD, Study Director — RTI International
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - RTI International, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Univeristy of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share IPD

REFERENCES:
- [Derived] Merhar SL, Bann CM, Mack N, Newman JE, Limperopoulos C, Ambalavanan N, Davis JM, DeMauro SB, Lorch SA, Wilson-Costello DE, Peralta-Carcelan M, Parlberg LM, Poindexter BB, Kapse K, Kline-Fath BM, Murnick JG. Prenatal Opioid Exposure Is Associated with Punctate White Matter Lesions in Term Newborns. J Pediatr. 2025 Sep;284:114669. doi: 10.1016/j.jpeds.2025.114669. Epub 2025 May 23. PMID 40414418
- [Derived] Wu Y, Merhar SL, Bann CM, Newman JE, Kapse K, De Asis-Cruz J, Mack N, De Mauro SB, Ambalavanan N, Davis JM, Lorch SA, Wilson-Costello D, Poindexter BB, Peralta-Carcelen M, Limperopoulos C. Antenatal Opioid Exposure and Global and Regional Brain Volumes in Newborns. JAMA Pediatr. 2025 Jun 1;179(6):639-646. doi: 10.1001/jamapediatrics.2025.0277. PMID 40193106
- [Derived] Parlberg LM, Newman JE, Merhar SL, Poindexter B, DeMauro SB, Lorch SA, Peralta-Carcelen M, Wilson-Costello DE, Ambalavanan N, Limperopoulos C, Mack N, Davis JM, Walsh MC, Bann CM; ACT NOW OBOE Study Consortium. Risk factors for food insecurity and association with prenatal care utilization among women who took opioids during pregnancy and unexposed controls. BMC Pregnancy Childbirth. 2025 Apr 4;25(1):396. doi: 10.1186/s12884-025-07499-y. PMID 40186111
- [Derived] Merhar SL, Yolton K, DeMauro SB, Beiersdorfer T, Newman JE, Lorch SA, Wilson-Costello D, Ambalavanan N, Bangdiwala A, Peralta-Carcelen M, Poindexter BB, Davis JM, Limperopoulos C, Bann CM. Neurobehavioral Profiles in Opioid-Exposed and Unexposed Neonates. J Pediatr. 2025 Jun;281:114527. doi: 10.1016/j.jpeds.2025.114527. Epub 2025 Mar 7. PMID 40057022
- [Derived] Parlberg LM, Newman JE, Merhar S, Poindexter B, DeMauro S, Lorch S, Peralta-Carcelen M, Wilson-Costello D, Ambalavanan N, Limperopoulos C, Mack N, Davis JM, Walsh M, Bann CM. Risk factors for food insecurity and association with prenatal care utilization among women who took opioids during pregnancy. Res Sq [Preprint]. 2024 Mar 25:rs.3.rs-3921909. doi: 10.21203/rs.3.rs-3921909/v1. PMID 38585728